CLINICAL TRIAL: NCT03641573
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C] ASN002 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Phase 1 Study to Evaluate ASN002 Absorption, Metabolism, and Excretion of [14C] Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASN002AD-102
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gusacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] ASN002 (Experimental): [14C] ASN002
  Interventions: Drug: [14C] ASN002

INTERVENTIONS:
Drug: [14C] ASN002 — [14C] ASN002

SUMMARY:
Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C] ASN002 Following a Single Oral Dose in Healthy Male Subjects

DETAILED DESCRIPTION:
This will be a Phase 1, open-label, nonrandomized, single-dose study in healthy male subjects. Subjects will be admitted into the Clinical Research Unit (CRU) on Day 1 and be confined to the CRU until at least Day 7. On Day 1, subjects will receive a single oral dose of [14C] ASN002 at 60 mg containing approximately 300 μCi [14C] ASN002. Subjects will be discharged on Day 7 if the following discharge criteria are met: plasma radioactivity levels below the limit of quantitation for 2 consecutive collections, and ≥90% mass balance recovery, or ≤1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 3 consecutive 24 hour periods. If discharge criteria are not met by Day 7, subjects will remain in the CRU up to a maximum of Day 10.

ELIGIBILITY:
Inclusion Criteria:

* Males, of any race, between 20 and 60 years of age, inclusive, at Screening.
* Body mass index between 18.5 and 30.0 kg/m2, inclusive, at Screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check in as assessed by the Investigator (or designee).
* Males will agree to use contraception as defined in the Protocol body
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will not be allowed).
* History of alcoholism or drug/chemical abuse within 2 years prior to Check in.
* Consumption of alcohol from 72 hours prior to Check-in until Discharge.
* Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges from 7 days prior to Check-in until Discharge.
* Consumption of caffeine containing foods and beverages from 48 hours before Check-in until Discharge.
* Positive urine drug screen (including cotinine) at Screening or positive alcohol breath test or positive urine drug screen (including cotinine) at Check in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known), whichever is longer, prior to Check-in.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or excretion processes, including St. John's wort, within 14 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any prescription medications/products within 14 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use slow release medications/products considered to still be active within 14 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
* Use of tobacco or nicotine containing products within 3 months prior to Check in.
* Receipt of blood products within 2 months prior to Check in.
* Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or any other study investigating ASN002, and have previously received the investigational medicinal product (IMP).
* Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
* Subjects who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study. The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the CFR recommended levels considered safe, per United States Title 21 CFR 361.1: less than 5,000 mrem whole body annual exposure with consideration given to the half-lives of the previous radiolabeled study drugs received.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Cmax - maximum observed plasma concentration (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
tmax - time at which Cmax occurs (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
AUC0 t - area under the plasma concentration time curve from time zero to the last measurable concentration (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
AUC0-∞ - area under the plasma concentration-time curve from time zero to infinity (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
t½ - apparent terminal elimination half-life (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
CL/F - apparent total clearance (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
VZ/F - apparent volume of distribution (plasma and whole blood) | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
Total radioactivity in urine and feces | at pre-dose and up to 144 hours post-dose. If collection is extended up to Day 10: at up to 216 hours post-dose.
  %Ae (urine), %Ae (feces) and %Ae (total): amount excreted and cumulative amount excreted in urine and feces

SECONDARY OUTCOMES:
Metabolic Profiling/identification and determination of relative abundance of ASN002 and the metabolites of ASN002 in plasma, urine, and feces | Up to 10 days
Safety and tolerability as measured by incidence and severity of adverse events (AEs) | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Niranjan Rao, PhD, Study Director — Asana BioSciences
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No